CLINICAL TRIAL: NCT03877887
Title: Comparison of Treatment and Doses of Drugs in Patient With Heart Failure Reduced Ejection Fraction (HFREF) Between Asyut University Hospital and Guidelines of European Society 0f Cardiology (ESC)
Brief Title: Finding Gab in the Treatment of Heart Failure in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Shnouda Halim, Principal investigator, Assiut University
Other Study IDs: heart failure in Assuit
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: echo cardiogram — Assessment of left ventricular systolic and diastolic function

SUMMARY:
Analyze the epidemiology and outcome of all patients with heart failure with reduced ejection fraction (HFrEF) presented to Asyut university hospital (AUH) and to identify factors associated with mortality and all-cause hospitalization at a duration of 6 months follow-up.

DETAILED DESCRIPTION:
Heart failure (HF) is nowadays an important health problem and associated with high use of resources and healthcare cost, but the prevalence of heart failure is increasing due to better care and treatment of HF and to the aging of the population. Epidemiology of HF is changing and shifting towards a higher prevalence of patients with HF with preserved ejection fraction. Moreover, the outcome of HF is grim. The mortality rate is high and hospitalizations are frequent and associated with worse outcomes. The majority of studies that analyzed HF outcomes have focused on HF hospitalizations. However, in patients with HF, all-cause hospitalizations can affect up to 23-58% of the patients at 1-year follow-up and non-cardiovascular hospitalizations are associated with risk of subsequent mortality similar to cardiovascular hospitalizations. Despite the evidence that all-cause hospitalizations are detrimental in HF patients, few studies have analyzed whether the factors associated with all-cause and HF-hospitalizations are different in HF patients.

However, the characteristics and outcome of HF patients are not well described in developing countries like Egypt. Documenting patients' characteristics and the outcome might improve management of comorbidities associated with heart failure patients in Egypt as well as the disease outcome, However, characteristics and outcome of HF patients are not well described in developing countries like Egypt. Documenting patients' characteristics and the outcome might improve management of comorbidities associated with heart failure patients in Egypt as well as the disease outcome, However, characteristics and outcome of HF patients are not well described in developing countries like Egypt. Documenting patients' characteristics and the outcome might improve management of comorbidities associated with heart failure patients in Egypt as well as the disease outcome However, characteristics and outcome of HF patients are not well described in developing countries like Egypt. Documenting patients' characteristics and the outcome might improve the management of comorbidities associated with heart failure patients in Egypt as well as the disease outcome

ELIGIBILITY:
Inclusion Criteria:

- All patients > 18 years of age with left ventricular ejection fraction (LVEF) < 40 % with symptoms and signs of heart failure (according to ESC guidelines of acute and chronic heart failure 2016).

Exclusion Criteria:

* patients more than 80 years old

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presented to Assiut university hospital outpatient clinic, inpatient ward and CCU admission with heart failure reduced ejection fraction according to inclusion criteria for 6 months from March 2019 to August 2019.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
To find the percentage of patients treated at guidelines recommended doses | six months
  All patients presented to Assiut university hospital outpatient clinic, inpatient ward and CCU admission with heart failure reduced ejection fraction will be grouped according to Age ( Etiology,risk factors,severity of symptoms (according to NYHA score),hospitalizations , co-morbidity and treatment and doses they received and compare it to guidelines and follow for re-hospitalization and mortality.

REFERENCES:
- [Background] Farre N, Vela E, Cleries M, Bustins M, Cainzos-Achirica M, Enjuanes C, Moliner P, Ruiz S, Verdu-Rotellar JM, Comin-Colet J. Real world heart failure epidemiology and outcome: A population-based analysis of 88,195 patients. PLoS One. 2017 Feb 24;12(2):e0172745. doi: 10.1371/journal.pone.0172745. eCollection 2017. PMID 28235067